CLINICAL TRIAL: NCT05173493
Title: The Study About the Selection of Time for Retreatment of Helicobacter Pylori After Eradication Failure
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Collaborators: Taian City Central Hospital (Other); Dezhou People's Hospital (Other); Weifang Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Shengli Oilfield Hospital (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Professor, Director of gastroenterology department of Qilu hospita, Shandong University
Other Study IDs: 2021-SDU-QILU-G101
Record Dates: First submitted 2021-12-28; First posted 2021-12-30 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Re-eradication time; Remedial treatment
MeSH Terms: interventions — Amoxicillin; Furazolidone; Levofloxacin; Tetracycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Amoxicillin-Furazolidone-containing quadruple group: Patients in amoxicillin-furazolidone-containing quadruple group will receive esomeprazole (Nexium) 40mg po bid(or vonoprazan fumarate 20mg po bid), amoxicillin1000mg po bid, bismuth potassium citrate(Lizhudele) 220mg po bid, and furazolidone (Liteling) 100mg po bid for 14d.
  Interventions: Drug: Amoxicillin,Furazolidone
- Amoxicillin-Levofloxacin-containing quadruple group: Patients in amoxicillin-Levofloxacin-containing quadruple group will receive esomeprazole (Nexium) 40mg po bid(or vonoprazan fumarate 20mg po bid), amoxicillin1000mg po bid, bismuth potassium citrate(Lizhudele) 220mg po bid, and levofloxacin 500mg po qd for 14d.
  Interventions: Drug: Amoxicillin,Levofloxacin
- Tetracycline-Furazolidone-containing quadruple group: Patients in tetracycline-furazolidone-containing quadruple group will receive esomeprazole (Nexium) 40mg po bid(or vonoprazan fumarate 20mg po bid), tetracycline 500 mg po qid, bismuth potassium citrate(Lizhudele) 220mg po bid, and furazolidone (Liteling) 100mg po bid for 14d.
  Interventions: Drug: Tetracycline,Furazolidone

INTERVENTIONS:
Drug: Amoxicillin,Furazolidone — Amoxicillin-Furazolidone-containing quadruple group
  Groups: Amoxicillin-Furazolidone-containing quadruple group
Drug: Amoxicillin,Levofloxacin — Amoxicillin-Levofloxacin-containing quadruple group
  Groups: Amoxicillin-Levofloxacin-containing quadruple group
Drug: Tetracycline,Furazolidone — Tetracycline-Furazolidone-containing quadruple group
  Groups: Tetracycline-Furazolidone-containing quadruple group

SUMMARY:
The patients who accepted the quadruple eradication program of the helicobacter pylori but failed to eradicate helicobacter pylori will be assessed the most suitable re-eradication time of helicobacter pylori.

DETAILED DESCRIPTION:
Helicobacter pylori (HP) infection is a common global infectious disease, which is an important cause of chronic gastritis, peptic ulcer and gastric cancer. At present, due to the non-standard Helicobacter pylori eradication program in clinical work, poor patient compliance and other reasons, the phenomenon of HP eradication treatment failure is more and more common. However, there is still no conclusion on the most appropriate time for remedial treatment inpatients with Hp eradication failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 with H. pylori infection.
* Patients with previous Helicobacter pylori eradication.

Exclusion Criteria:

* Patients treated with H2-receptor antagonist, PPI, bismuth and antibioticsin the previous 4 weeks.
* Patients with gastrectomy, acute GI bleeding and advanced gastric cancer.
* Patients with known or suspected allergy to study medications.
* Currently pregnant or lactating.
* Inability to provide informed consent and other situations that couldinterfere with the examination or therapeutic protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients in Shandong province,aged between 18 and 70 years old, with positive H. pylori infection that was eradicated by previous therapies but failed are included.
Sampling Method: Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
The most suitable re-eradication time | 6 months
  The most suitable re-eradication time（The unit is month） will be assessed by paired comparison method .

SECONDARY OUTCOMES:
Eradication rates in three groups | 6months
  Both intention to treat(ITT) and per-protocol(PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Lin M, Hu J, Liu J, Wang J, Han Z, Wang X, Zhai Z, Yu Y, Yuan W, Zhang W, Wang Z, Kong Q, Lin B, Ding Y, Wan M, Zhang W, Duan M, Zeng S, Li Y, Zuo X, Li Y. The interval of rescue treatment does not affect the efficacy and safety of Helicobacter pylori eradication: A prospective multicenter observational study. Chin Med J (Engl). 2025 Jun 20;138(12):1439-1446. doi: 10.1097/CM9.0000000000003534. Epub 2025 Apr 29. PMID 40304303